CLINICAL TRIAL: NCT03085979
Title: Surgical Management of Mixed Urinary Incontinence
Brief Title: Mixed Urinary Incontinence Surgical Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams Maternity Hospital (Other)
Responsible Party: Principal Investigator, Hamdy Ahmed Saaid, Fellow of OBSlGYN, Ain Shams Maternity Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MUIT
Record Dates: First submitted 2017-03-10; First posted 2017-03-22 (Actual); Last update posted 2022-07-27 (Actual); Status verified 2022-07

CONDITIONS: Med: Urinary Incontinence (Stress, Urge, Mixed)
MeSH Terms: interventions — Suburethral Slings

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Burch (Experimental): Burch Colposuspension
  Interventions: Procedure: Burch Colposuspension
- Trans Obturator Tape (Experimental): Trans Obturator Tape sling
  Interventions: Procedure: trans obturator tape
- Tension free vaginal tape (Experimental): Tension free vaginal tape sling
  Interventions: Procedure: tension free vaginal tape

INTERVENTIONS:
Procedure: Burch Colposuspension — Anti-incontinent surgery
  Arms: Burch
Procedure: trans obturator tape — Anti-incontinent surgery
  Arms: Trans Obturator Tape
Procedure: tension free vaginal tape — Anti-incontinent surgery
  Arms: Tension free vaginal tape

SUMMARY:
Surgical management of mixed urinary incontinence

DETAILED DESCRIPTION:
Study to evaluate role of anti-incontinent surgery Burch colposuspension Tension free vaginal tape Trans obturator tape for the management of mixed urinary incontinence .

ELIGIBILITY:
Inclusion Criteria:

* patients with Mixed urinary incontinence

Exclusion Criteria:

Women with associated gynecological surgery e.g. uterine prolapse, previous anti-incontinence surgery, intrinsic sphincter deficiency (ISD), and medical disorders affecting the bladder innervation as diabetes mellitus were excluded from the study. Women who improved on medical treatment with persistence of stress element only were also excluded.

Ages: 20 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 198 (Actual)
Dates: Start 2014-10 (Actual); Primary Completion 2018-10 (Actual); Study Completion 2022-05 (Actual)

PRIMARY OUTCOMES:
cure of Mixed incontinence | 1 year
  compare the 3 groups as regard cure rate of both Components of mixed incontinence

CONTACTS AND LOCATIONS:
Overall Officials: Hamdy HA Ahmed Saaid, M.D, Principal Investigator — Fellow of OBS/GYN

IPD SHARING:
Plan to Share IPD: No